CLINICAL TRIAL: NCT01292967
Title: The Influence of Maltitol on the Absorption and Metabolism of Flavanols From Chocolate
Brief Title: Influence of Sugar on the Bioavailability of Cocoa Flavanols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Dr Jeremy P E Spencer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UReading-2010_03
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Flavanol; cocoa; maltitol; absorption; metabolism; chocolate; food matrix; bioavailability
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low flavanol (Placebo Comparator): Low-flavanol chocolate contained 48 mg of cocoa flavanols. macro- and micro-nutrient matched with active comparator
  Interventions: Dietary Supplement: Low flavanol chocolate
- High-flavanol with sugar (Active Comparator): High-flavanol chocolate made with added sugar containing 251 mg of cocoa flavanols
  Interventions: Dietary Supplement: High-flavanol with sugar
- High flavanol Maltitol (Active Comparator): High-flavanol chocolate made with the sugar substitute maltitol containing 266 mg cocoa flavanols
  Interventions: Dietary Supplement: High flavanol Maltitol

INTERVENTIONS:
Dietary Supplement: Low flavanol chocolate — 48 mg of total flavanols from cocoa
  Arms: Low flavanol
Dietary Supplement: High-flavanol with sugar — high-flavanol containing 251 mg cocoa flavanols
  Arms: High-flavanol with sugar
Dietary Supplement: High flavanol Maltitol — high-flavanol containing 266 mg cocoa flavanols
  Arms: High flavanol Maltitol

SUMMARY:
The primary propose of this study is to determine the impact of ingredients and matrices on flavanol absorption and metabolism.

DETAILED DESCRIPTION:
The investigators have conducted a randomized, triple-blind, cross-over study in 15 healthy human volunteers to investigate the absorption and metabolism of cocoa flavanols from a high-flavanol chocolate made with added sugar and a high-flavanol chocolate containing the sugar substitute maltitol; a nutrient-matched low flavanol control product was also fed. All products were matched for macro-nutrients, as well as for alkaloids (theobromine and caffeine), and were similar in taste and appearance. Both high-flavanol products contained ~259 mg cocoa flavanols, whilst the low-flavanol chocolate contained 48 mg of cocoa flavanols. On each study day, subjects were cannulated and baseline blood samples were collected prior to consumption of any of the test chocolates. Additional blood samples were collected at 1, 2 and 4 hours and plasma levels of flavanols were assessed using HPLC with fluorescence detection. All test products were well-tolerated by study participants.

ELIGIBILITY:
Inclusion Criteria:

* a signed consent form
* age of 18-50 years inclusive

Exclusion Criteria:

* did not suffer from any form of disease, including liver disease, diabetes mellitus or a myocardial infarction
* not on medications for the treatment of hypertension, elevated lipids or diabetes (type I and II).
* did not suffered gall bladder problems or abnormalities of fat metabolism
* weight reducing dietary regimen or taking any dietary supplements, including dietary fatty acids
* did not consume more than 15 units (120g) of alcohol per week
* did not have sensitivities to chocolate, reduced calorie sweeteners, dairy, nuts or gluten.
* Vegetarians and vegans
* taken antibiotics in the last 8 weeks

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Impact of ingredients and matrices on flavanol absorption and metabolism. | 4 hours
  The absorption and metabolism of cocoa flavanols from a high-flavanol chocolate made with added sugar and a high-flavanol chocolate containing the sugar substitute maltitol will be assessed by using HPLC with fluorescence detection

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom